CLINICAL TRIAL: NCT02553785
Title: Clinical Study of the BioVentrix Revivent TC for the Treatment of Ischemic Cardiomyopathy
Acronym: ReviventTC1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVentrix (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0056
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: BioVentrix; Revivent; Revivent TC
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revivent TC (Experimental): Surgical treatment of left ventricle using the Revivent TC System
  Interventions: Device: Revivent TC

INTERVENTIONS:
Device: Revivent TC

SUMMARY:
This study is a multi-center, prospective, single-armed, study designed to evaluate the safety and efficacy of the BioVentrix Revivent TransCatheter (TC) System for left ventricular (LV) volume reduction in heart failure (HF).

DETAILED DESCRIPTION:
The purpose of this prospective, single-armed, multi-center clinical trial is to further establish the feasibility of using the BioVentrix Revivent TC System for the treatment of left ventricular dysfunction in appropriate cohorts of humans suffering from heart failure.

The objective of this study is to determine the safety and functionality of a device that enables left ventricle (LV) volume and radius reduction through scar exclusion in appropriate patients suffering from systolic HF. Use of this device replicates the geometric reconfiguration of the ventricle achieved through surgical Left Ventricular Reconstruction (LVR), but on a beating heart, and creates the option of eliminating the use of Cardiopulmonary Bypass.

The System utilizes anchors that are implanted into the scarred portion of the heart, rendering the ventricle smaller, and is employed in a cardiac surgical setting without the use of cardiopulmonary bypass. The Revivent TC anchors may be implanted through a sternotomy or through a mini-thoracotomy and jugular access. Eligible subjects will be limited to those whose ventricular dysfunction is due to ischemic cardiomyopathy caused, by a previous (greater than 90 days) myocardial infarction (MI) with acontractile (akinetic and/or dyskinetic) scar located in the antero-septal, apical (may extend laterally) region.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80;
* Left Ventricular Ejection Fraction (LVEF) >15% and ≤ 45%;
* New York Heart Association (NYHA) Functional Class II-IV;
* Left Ventricular End Systolic Volume (LVESVI) ≥60 cc/m² but ≤ 120 cc/ m²
* Contiguous acontractile (akinetic and/or dyskinetic) scar located in the antero-septal, apical (may extend laterally) regions of the left ventricle as evidenced by a Cardiac Magnetic Resonance (CMR) or Computed Tomography (CT);
* Maintained standard medical management for at least 90 days, and at stable target (or maximum tolerated) dosages;
* Willing and competent to complete informed consent;
* Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by CMR or CT;
* Agree to required follow-up visits

Exclusion Criteria:

* Calcified ventricular wall in the area of intended scar exclusion as verified by echocardiography or equivalent;
* Thrombus or intra-ventricular mass in the left atrium or ventricle as verified by echocardiography or equivalent;
* Cardiac Resynchronization Therapy (CRT) device placement ≤ 60 days prior to enrollment;
* Significant diastolic dysfunction, defined as a pseudo-normal Doppler filling pattern with E/A ratio > 2;
* Thin walled, paradoxically moving septal scar that would preclude successful support of the anchor pairs as evidenced by CMR;
* Cardiac valve disease which, in the opinion of the investigator, will require surgery;
* Intolerance or unwillingness to take anti-coagulation medication;
* Functioning pacemaker leads in antero-apical right ventricle, which, in the opinion of the investigator, would interfere with anchor placement;
* Pulmonary Arterial Pressure > 60 mm Hg via echo;
* Myocardial Infarction within 90 days prior to enrollment;
* Previous Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) which resulted, in the opinion of the investigator, in a significant residual neurological deficit;
* Aorto iliac disease that would preclude fem-fem bypass.
* Previous right neck surgery, previous pericardiotomy, previous left chest surgery;
* Co-morbid disease process with life expectancy of less than one year;
* Patients with lung, kidney and/or liver transplant;
* Chronic renal failure with a serum creatinine >2 mg/dL;
* Inoperable coronary disease with significant ischemia;
* Pregnant or planning to become pregnant during the study;
* Enrolled in any concurrent study other than observational.
* Previous left thoracotomy
* Pulmonary disease that would preclude single lung ventilation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 6 months
  Overall rate of serious adverse events (SAEs)
Primary Efficacy Endpoint | 6 months
  Decrease in LV volume (left ventricular end-systolic volume index) compared to Baseline

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 6 months
  Rate of Serious Adverse Device Effects
Secondary Efficacy Endpoint | 6 months
  Change in Left Ventricular Ejection Fraction compared to Baseline
Secondary Efficacy Endpoint | 6 months
  Hospital readmission for Heart Failure
Secondary Efficacy Endpoint | 6 months
  Change in NYHA failure class compared to Baseline
Secondary Efficacy Endpoint | 6 months
  Change in a standardized 6-minute corridor walk test compared to Baseline
Secondary Efficacy Endpoint | 6 months
  Change in Quality of Life (QOL) by Minnesota Living with Heart Failure (MLHF) Questionnaire compared to Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic University of Barcelona, Barcelona, Spain

REFERENCES:
- See also: Sponsor Website — http://www.bioventrix.com